CLINICAL TRIAL: NCT06374862
Title: Effects of Specific Thoracic Spine Mobilizations on Muscle Activity in a Healthy Volunteer Population
Acronym: RACHIMOB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PI2024_843_0008
Record Dates: First submitted 2024-04-16; First posted 2024-04-19 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Musculoskeletal Manipulations; Range of Motion; Muscle Strength; Peripheral Joints in Upper Quarters
Keywords: Musculoskeletal Manipulations; Range of Motion; Muscle Strength; peripheral joints in upper quarters
MeSH Terms: interventions — No-Observed-Adverse-Effect Level

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Interventional (Experimental): This study is of an interventional nature, because the investigators want to objectively assess the impact of specific mobilization on neuromuscular functioning, thanks to surface EMG, before and after a specific mobilization of the spine.
  Interventions: Other: mobilization
- control (Sham Comparator): This approach will help to determine whether there is spontaneous modulation of neuromuscular activity in the absence of intervention. Thus, the investigators can distinguish the effects of intervention from natural variations in the healthy subject.
  Interventions: Other: no effect
- no interventional (No Intervention): A control group was also integrated to assess whether a mobilization identified as "no effect" could modulate neuromuscular activity by a placebo effect. This approach will allow to disentangle the real effects of mobilization from those that could result from psychomotor responses

INTERVENTIONS:
Other: mobilization — specific mobilization on neuromuscular functioning, thanks to surface EMG, before and after a specific mobilization of the spine
  Arms: Interventional
Other: no effect — a mobilization identified as "no effect" could modulate neuromuscular activity by a placebo effect.
  Arms: control

SUMMARY:
In this study, the investigators will examine the effect of manual therapy on the thoracic spine and its impact on the muscular strength gain of the thoracic extensors. Treatment with manual therapy, as described by Maitland, consists of a specific mobilization of the thoracic spine in the postero-anterior direction on the transverse and spiny processes of the thoracic vertebrae. To ensure the relevance of the measures, and to better control the occurrence of biases inherent to the practice of manual therapy, the investigators constituted three distinct groups: an intervention group, a control group and a group without intervention. In short, this methodology will allow us to explore in detail the effects of specific spinal mobilization on motor control, while taking into account placebo response elements and natural variations in the results

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 to 65,
* healthy volunteer,
* membership in a social security scheme

Exclusion Criteria:

* Severe spinal trauma within the last 6 months
* history of low back pain, back pain, and/or neck pain within the last 6 months,
* history of spinal surgery,
* history of chronic systemic disease (cardiac, respiratory, diabetes, etc.),
* volunteer with Pacemaker, history of rheumatological pathology (rheumatoid arthritis, ankylosing spondylitis, Scheuermann's disease, etc.),
* patient under guardianship,curatorship, safeguard of justice, patient deprived of liberty, pregnant woman and patient without Red Flags Social Security described in literature.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2024-03-28 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
electrical activity assessment of the spine extensor muscles using EMG | 1 hour

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, Picardie, France

IPD SHARING:
Plan to Share IPD: No